CLINICAL TRIAL: NCT00390429
Title: Phase I/II Study of Docetaxel and OSI-774 (Erlotinib) in Solid Tumor Patients With an Emphasis on NSCLC Using Molecular Correlates as Potential Markers of Response
Brief Title: Docetaxel and Erlotinib in Treating Patients With Advanced Non-Small Cell Lung Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 273721; P30CA093373 (NIH); UCDCC-128 (Other: University of California, Davis - Cancer Center); UCDCC-200311717-5 (Other: University of California, Davis - IRB); AVENTIS-Z1001055 (Other: Aventis Pharmaceuticals); CDR0000505821 (Other: UC Davis)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I, Group I (completed) (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib hydrochloride once on days 2, 9, and 16. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: docetaxel; Drug: erlotinib hydrochloride
- Phase I, Group II (completed) (Experimental): Patients receive docetaxel as in group I and oral erlotinib hydrochloride once daily on days 2-16. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: docetaxel; Drug: erlotinib hydrochloride
- Phase II (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib hydrochloride at the MTD determined in group II of phase I once daily on days 2-16. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may then continue to receive erlotinib hydrochloride alone in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: Taxotere
Drug: erlotinib hydrochloride — Given orally
  Other Names: OSI-774; Tarceva

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving docetaxel together with erlotinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of erlotinib when given together with docetaxel in treating patients with solid tumors and to see how well they work in treating patients with advanced non-small cell lung cancer. (Phase I portion of the study treating patients with any solid tumor was completed as of 12/01/2004)

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of two different schedules of erlotinib hydrochloride and docetaxel in patients with advanced solid tumors. (Phase I [completed as of 12/01/2004])
* Determine the response rate in patients with advanced non-small cell lung cancer treated with second-line docetaxel and erlotinib hydrochloride. (Phase II)

Secondary

* Compare the toxicity of two different schedules of erlotinib hydrochloride and docetaxel in these patients. (Phase I [completed as of 12/01/2004])
* Determine the maximum tolerated dose of two different schedules of erlotinib hydrochloride and docetaxel. (Phase I [completed as of 12/01/2004])
* Assess the overall survival and progression-free survival. (Phase II)
* Determine the frequency and severity of toxicities associated with this treatment regimen. (Phase II)

Tertiary

* Perform laboratory correlative studies on patient tissue and blood samples to investigate potential predictors of response.

OUTLINE: This is a phase I, dose-escalation study of erlotinib hydrochloride (phase I completed as of 12/01/2004) followed by a phase II, open-label study.

* Phase I (completed as of 12/01/2004): Patients will be assigned in alternating fashion to 1 of 2 treatment groups.

  * Group I: Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib hydrochloride once on days 2, 9, and 16.
  * Group II: Patients receive docetaxel as in group I and oral erlotinib hydrochloride once daily on days 2-16.

In both groups, treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.

In both groups, cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib hydrochloride at the MTD determined in group II of phase I once daily on days 2-16. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may then continue to receive erlotinib hydrochloride alone in the absence of disease progression or unacceptable toxicity.

Blood samples, buccal mucosal cells, and tumor tissue are obtained before and after treatment. Epidermal growth factor receptor (EGFR) expression and polymorphisms and p27 protein expression are assessed by immunohistochemistry. Immunofluorescence (by laser-scanning cytometry) is used to detect EGFR and p27.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 87 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* For the phase II portion patients must have cytologically or histologically proven NSCLC. (Completed 12/1/04 - For the phase I portion of the study patients must have cytologically or histologically proven advanced solid tumors for which there is no standard therapy of curative intent).
* For the phase II portion patients must have disease that has progressed or recurred after treatment with platinum based therapy. Patients that have stable disease after front line platinum based therapy is also eligible.
* No more than 1 previous treatment for metastatic disease is allowed for the phase II portion. (Completed 12/1/04 - Any number of prior chemotherapy regimens for metastatic disease are allowed for the phase I portion).
* Patients must have measurable disease by RECIST criteria. Disease in previously irradiated sites is considered measurable if there is clear disease progression following radiation therapy. (Completed 12/1/04 - Patients with evaluable disease may be included in the phase I portion of the trial.
* Patients must be 18 years of age or older.
* Patients must have a performance status of 0-1 for the phase II portion of the trial. (Completed 12/1/04 - performance status of 0-2 for is allowed for the phase I portion of study
* Patients must have an estimated survival of at least 3 months.
* Any prior chemotherapy that patients have received has to have been completed at least 4 weeks prior to start of OSI-774/Docetaxel. For prior mitomycin chemotherapy a 6-week interval is required. Prior radiation must have been completed at least 2 weeks prior to start of therapy. All side effects must have resolved prior to start of OSI-774/Docetaxel.
* Patients must have adequate renal function as documented by a serum creatinine < 1.5 mg/dl or a calculated creatinine clearance of > 50 ml/min (see appendix for formula for calculating creatinine clearance).
* Patients must have adequate liver function as documented by serum bilirubin < ULN. AST must be < 2.5 x institutional upper limit of normal.
* Patients must have a pretreatment granulocyte count of >1500/mm3 and platelet count of >100 000/mm3.
* Patients with asymptomatic treated brain metastasis (surgical resection or radiotherapy) may be included if they are neurologically stable and have been off steroids and anticonvulsants for at least 4 weeks. Because of the possibility of treatment related neurological toxicity it is difficult to evaluate for toxicity in the presence of symptomatic brain metastasis.
* All patients must give written informed consent.
* Able to take and retain oral medication.
* Patients of reproductive potential must agree to use effective contraceptive method while on treatment and for 3 months afterwards as the effects of these drugs on the unborn fetus are unknown.
* Patients on Coumadin should have their INR monitored at least once per week or more frequently depending on the investigators judgment. There have been some case reports of increased INR when Coumadin is co-administered with OSI-774/placebo.

Exclusion Criteria:

* May not have previously received docetaxel; OSI-774 or any prior EGFR targeted therapy.
* Females can not be pregnant or breastfeeding as the effects of these drugs on the unborn fetus are unknown. Documentation of a negative pregnancy test is required for all women of reproductive potential.
* Patients with symptomatic brain metastasis or still requiring steroids may not be included.
* Clinically significant ophthalmologic abnormalities will be excluded. This includes severe dry eye syndrome, keratoconjunctivitis sicca, Sjogren's syndrome, severe exposure keratopathy, or other disorders that might increase the risk of corneal epithelial injury.
* A history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* Pre-existing neuropathy > grade 2 may not participate
* No other prior malignancy is allowed for the phase II portion except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for over five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2002-07; Primary Completion 2008-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Gandara, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Group A (1200 mg Erlotinib + 70mg/m2 Docetaxel): Original Dose Level
  Patients receive docetaxel IV over 1 hour on day 1 and oral Erlotinib hydrochloride once on days 2, 9, and 16 and Docetaxel on days 1 and 22. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  Docetaxel: Given IV Erlotinib hydrochloride: Given orally
- Phase I, Group A (600 mg Erlotinib + 70mg/m2 Docetaxel): Patients receive docetaxel IV over 1 hour on day 1 and oral Erlotinib hydrochloride once on days 2, 9, and 16 and Docetaxel on days 1 and 22. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  Docetaxel: Given IV Erlotinib hydrochloride: Given orally
- Phase I, Group B (Completed): Patients receive docetaxel as in group I and oral erlotinib hydrochloride once daily on days 2-16. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  docetaxel: Given IV erlotinib hydrochloride: Given orally
- Phase II: Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib hydrochloride at the MTD determined in group II of phase I once daily on days 2-16. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may then continue to receive erlotinib hydrochloride alone in the absence of disease progression or unacceptable toxicity.
  docetaxel: Given IV erlotinib hydrochloride: Given orally
Period: Overall Study
Arm/Group | Phase I, Group A (1200 mg Erlotinib + 70mg/m2 Docetaxel) | Phase I, Group A (600 mg Erlotinib + 70mg/m2 Docetaxel) | Phase I, Group B (Completed) | Phase II
Started | 5 | 12 | 25 | 39
Completed | 5 | 12 | 25 | 39
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I, Arm A (Completed): Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib hydrochloride once on days 2, 9, and 16. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  docetaxel: Given IV
  erlotinib hydrochloride: Given orally
- Phase I, Arm B (Completed): Patients receive docetaxel as in group I and oral erlotinib hydrochloride once daily on days 2-16. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  docetaxel: Given IV
  erlotinib hydrochloride: Given orally
- Total: Total of all reporting groups
Arm/Group | Phase I, Arm A (Completed) | Phase I, Arm B (Completed) | Phase II | Total
Number analyzed (Participants) | 17 | 25 | 39 | 81
Age, Continuous [Median (Full Range); unit: years] | 63 [40 to 75] | 55 [34 to 83] | 61 [38 to 80] | 61 [34 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 24 | 44
  Male | 11 | 11 | 15 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African descent | 1 | 0 | 2 | 3
  Race: White | 15 | 23 | 35 | 73
  Race: East/South East Asian | 1 | 2 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 17 | 25 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Safety and Toxicity of Erlotinib Hydrochloride and Docetaxel as Measured by NCI CTC v3.0 on Day 8 of Course 1 and on Day 1 of Every Subsequent Course (Phase I [Completed as of 12/01/2004])
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Arm A (Completed) | Phase I, Arm B (Completed) | Phase II
Number analyzed (Participants) | 17 | 25 | 39
Participants | 17 | 25 | 39

2. Primary Outcome: Response Rate (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 36 months
Population: All participants for whom response evaluation measurements were recorded at Baseline and after 2 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II
Number analyzed (Participants) | 39
Participants | 11

3. Secondary Outcome: Comparison of Toxicity of Two Different Schedules of Erlotinib Hydrochloride and Docetaxel (Phase I [Completed as of 12/01/2004])
Time Frame: up to 36 months
Measure: Number; unit: participants
Groups:
- Phase I, Group A (Completed): Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib hydrochloride once on days 2, 9, and 16. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients may then continue to receive erlotinib hydrochloride alone in the absence of unacceptable toxicity or disease progression.
  docetaxel: Given IV erlotinib hydrochloride: Given orally
Arm/Group | Phase I, Group A (Completed) | Phase I, Group B (Completed)
Number analyzed (Participants) | 17 | 25
participants
  Neutropenia | 10 | 16
  Febrile neutropenia | 3 | 4
  Hemoglobin | 0 | 1
  Diarrhea | 0 | 3
  Fatigue | 0 | 1
  Infection (without neutropenia) | 1 | 3
  Mucositis | 0 | 1
  Nausea | 1 | 0
  Rash | 0 | 1

4. Secondary Outcome: Maximum Tolerated Dose of Two Different Schedules of Erlotinib Hydrochloride and Docetaxel (Phase I [Completed as of 12/01/2004])
Description: Maximum tolerated dose (MTD) defined as the highest dose level at which no more than one patient experienced DLT when at least 6 patients were treated at that dose level and were assessable for toxicity, graded according to NCI CTCAE 2.0.
Time Frame: up to 36 months
Population: Phase I, arm A, MTD: erlotinib 600-1000 mg d 2, 9, and 16; and docetaxel 70 mg/m^2 d 1 on a 21-d cycle.
  Phase I, arm B, MTD: erlotinib 150-300 mg d 2 and 16; and docetaxel 70 mg/m^2 d 1 on a 21-d cycle.
Measure: Number; unit: mg
Arm/Group | Phase I, Group A (Completed) | Phase I, Group B (Completed)
Number analyzed (Participants) | 12 | 25
mg | 600 | 200

5. Secondary Outcome: Overall Survival (Phase II)
Time Frame: Up to 65 months
Measure: Median (Full Range); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 39
months | 18.2 [0 to 65]

6. Secondary Outcome: Progression-free Survival (Phase II)
Time Frame: Completion of study (up to 65 months)
Measure: Median (Full Range); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 39
months | 4.1 [0 to 65]

7. Secondary Outcome: Frequency and Severity of Toxicities (Phase II)
Description: Treatment-related adverse events Grade ≥3 by NCI CTCAE 2.0.
Time Frame: Completion of study (up to 36 months)
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 39
participants
  Neutropenia | 14
  Febrile neutropenia | 4
  Platelets | 1
  Diarrhea | 7
  Dehydration | 2
  Fatigue | 2
  Hypokalemia | 1
  Hyponatremia | 1
  Infection (without neutropenia) | 1
  Myalgias | 1
  Nausea | 1
  Ocular | 1
  Pain | 1
  Stomatitis | 1

8. Secondary Outcome: Prognostic Significance of Epithelial Growth Factor Receptor (EGFR) Expression
Time Frame: Completion of study (up to 36 months)
Population: Data were not collected.
Arm/Group | Phase II
Number analyzed (Participants) | 0

9. Secondary Outcome: Correlation of Baseline EGFR Levels With Clinical Outcome
Time Frame: Completion of study (up to 36 months)
Population: Data were not collected.
Arm/Group | Phase II
Number analyzed (Participants) | 0

10. Secondary Outcome: Correlation of Basal Levels of p27 With Response Rate and Overall Survival
Time Frame: Completion of study (up to 36 months)
Population: Data were not collected.
Arm/Group | Phase II
Number analyzed (Participants) | 0

11. Secondary Outcome: Correlation of Phospho-EGFR With Increased p27 and Clinical Outcome
Time Frame: Completion of study
Population: Data were not collected.
Arm/Group | Phase II
Number analyzed (Participants) | 0

12. Secondary Outcome: Correlation of EGFR Polymorphisms With Treatment Response and Clinical Outcome
Time Frame: Completion of study
Population: Data were not collected.
Arm/Group | Phase II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Phase I, Arm A (Completed) | Phase I, Arm B (Completed) | Phase II
Serious Adverse Events (participants affected / at risk) | 2/17 | 5/25 | 1/39
Other Adverse Events (participants affected / at risk) | 15/17 | 25/25 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Arm A (Completed) (N=17) | Phase I, Arm B (Completed) (N=25) | Phase II (N=39)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukocytes (Blood and lymphatic system disorders) | 0 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 0
GI Bleed (Gastrointestinal disorders) | 0 | 1 | 0
Clinically Documented Infection (Infections and infestations) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Arm A (Completed) (N=17) | Phase I, Arm B (Completed) (N=25) | Phase II (N=39)
Neutropenia (Blood and lymphatic system disorders) | 10 | 16 | 14
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 4
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 0
Platelets (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 2
Infection (without neutropenia) (Infections and infestations) | 1 | 3 | 1
Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Myalgias (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ocular (Eye disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes